CLINICAL TRIAL: NCT01565889
Title: Part A: Drug Interaction Study Between GS-7977 and Antiretroviral Therapy (ARV) Combinations of Efavirenz, Tenofovir and Emtricitabine; Efavirenz, Zidovudine and Lamivudine; Atazanavir/Ritonavir, Tenofovir and Emtricitabine; Darunavir/Ritonavir, Tenofovir and Emtricitabine; Raltegravir, Tenofovir and Emtricitabine in Human Immunodeficiency Virus and Hepatitis C Virus (HIV/HCV) Co-infected Patients. Part B: A Phase 2, Open-Label Study to Investigate the Efficacy and Safety of GS-7977 With Peginterferon Alfa 2a and Ribavirin for 12 Weeks in Treatment-Naïve HIV/HCV Co-infected Patients.
Brief Title: Part A: Drug Interaction Study of Sofosbuvir and Antiretroviral Therapy (ART) Combinations in HIV and Hepatitis C Virus (HCV) Co-infected Patients. Part B: Efficacy and Safety of Sofosbuvir for 12 Weeks in HIV/HCV Co-infected Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P7977-1910
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; lamivudine, zidovudine drug combination; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: SOF+EFV/FTC/TDF (Cohort 1) (Experimental): Participants with a prestudy regimen of EFV/FTC/TDF will receive SOF+EFV/FTC/TDF FDC for 7 days, followed by EFV/FTC/TDF FDC (or EFV+FTC/TDF) for 7 days, coadministered once daily in the evening under fasting conditions.
  Interventions: Drug: SOF; Drug: EFV/FTC/TDF
- Part A: SOF+EFV+ZDV/3TC (Cohort 2) (Experimental): Participants with a prestudy regimen of EFV+ZDV/3TC will receive SOF+EFV+ZDV/3TC for 7 days followed by EFV+ZDV/3TC for 7 days. Sofosbuvir and EFV will be administered once daily in the evening under fasting conditions; ZDV/3TC will be administered twice daily, in the morning without regard to food and in the evening on an empty stomach.
  Interventions: Drug: SOF; Drug: EFV; Drug: ZDV/3TC
- Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) (Experimental): Participants with a prestudy regimen of RTV+ATV+FTC/TDF will receive SOF+RTV+ATV+FTC/TDF for 7 days followed by RTV+ATV+FTC/TDF for 7 days coadministered once daily in the morning with food.
  Interventions: Drug: SOF; Drug: ATV; Drug: Ritonavir; Drug: FTC/TDF
- Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) (Experimental): Participants with a prestudy regimen of RTV+DRV+FTC/TDF will receive SOF+RTV+DRV+FTC/TDF for 7 days followed by RTV+DRV+FTC/TDF for 7 days coadministered once daily in the morning with food.
  Interventions: Drug: SOF; Drug: Ritonavir; Drug: FTC/TDF; Drug: DRV
- Part A: SOF+RAL+FTC/TDF (Cohort 5) (Experimental): Participants with a prestudy regimen of RAL+FTC/TDF will receive SOF+RAL+FTC/TDF for 7 days followed by RAL+FTC/TDF for 7 days. Sofosbuvir and FTC/TDF will be administered once daily in the morning with food; RAL will be administered twice daily, in the morning with food and in the evening without regard to food.
  Interventions: Drug: SOF; Drug: FTC/TDF; Drug: RAL
- Part B: SOF+PEG+RBV (Experimental): Participants will receive SOF+PEG+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: PEG; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg (1 × 400 mg tablet or 2 × 200 mg tablets) administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: EFV/FTC/TDF — Efavirenz (EFV) 600 mg/emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg fixed-dose combination (FDC) tablet administered orally once daily
  Other Names: Atripla®
  Arms: Part A: SOF+EFV/FTC/TDF (Cohort 1)
Drug: EFV — Efavirenz (EFV) 600 mg tablet administered orally once daily
  Other Names: Sustiva®
  Arms: Part A: SOF+EFV+ZDV/3TC (Cohort 2)
Drug: ZDV/3TC — Zidovudine (ZDV) 300 mg/lamivudine (3TC) 150 mg FDC tablet administered orally twice daily
  Other Names: Combivir®
  Arms: Part A: SOF+EFV+ZDV/3TC (Cohort 2)
Drug: ATV — Atazanavir (ATV) 400 mg tablet administered orally once daily
  Arms: Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3)
Drug: Ritonavir — Ritonavir (RTV) 100 mg tablet administered orally once daily
  Arms: Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3); Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4)
Drug: FTC/TDF — FTC/TDF (200/300 mg) FDC tablet administered orally once daily
  Other Names: Truvada®
  Arms: Part A: SOF+RAL+FTC/TDF (Cohort 5); Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3); Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4)
Drug: DRV — Darunavir (DRV) 800 mg (2 × 400 mg tablets) administered orally once daily
  Arms: Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4)
Drug: RAL — Raltegravir (RAL) 400 mg administered administered orally twice daily
  Arms: Part A: SOF+RAL+FTC/TDF (Cohort 5)
Drug: PEG — Pegylated interferon alfa (PEG) 180 μg administered once weekly by subcutaneous injection
  Other Names: Pegasys®
  Arms: Part B: SOF+PEG+RBV
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
  Arms: Part B: SOF+PEG+RBV

SUMMARY:
This study consists of 2 parts, Part A and Part B. Part A, the Phase 1 drug interaction/early viral kinetic study, will evaluate the effect of selected antiretroviral therapies on the safety, viral kinetics, and pharmacokinetics of sofosbuvir (GS-7977; PSI-7977) and its metabolites in participants with HIV and hepatitis C virus (HCV) coinfection. Part B, the Phase 2 treatment study, will investigate the efficacy and safety of sofosbuvir, pegylated interferon alpha (PEG) and ribavirin (RBV) in participants with HIV/HCV coinfection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy according to medical history and physical examination with exception of HCV and HIV diagnoses
* Confirmation of Chronic HCV infection
* Confirmation of Chronic HIV-1 infection
* On a stable protocol approved HIV antiretroviral (ARV) regimen with undetectable HIV-RNA
* Agree to use two forms of highly effective contraception for the duration of the study and 6 months after the last dose of study medication
* Subjects must be naive to treatment for chronic HCV infection

Exclusion Criteria:

* Known or suspected cirrhosis
* History of any other clinically significant chronic liver disease
* A history consistent with decompensated liver disease.
* Use of any prohibited medications as defined by the protocol
* Pregnant or nursing female or male with pregnant female partner
* Contraindication to PEG or RBV therapy (for Part B)
* Clinically relevant drug or alcohol abuse

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Gaggar, MD/PhD, Study Director — Gilead Sciences
Locations (1):
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Rodriguez-Torres M, Gaggar A, Shen G, Kirby B, Svarovskaia E, Brainard D, Symonds WT, McHutchison JG, Gonzalez M, Rodriguez-Orengo J. Sofosbuvir for chronic hepatitis C virus infection genotype 1-4 in patients coinfected with HIV. J Acquir Immune Defic Syndr. 2015 Apr 15;68(5):543-9. doi: 10.1097/QAI.0000000000000516. PMID 25622055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 participants were enrolled at one study site in Puerto Rico, a commonwealth of the United States (US). The first participant was screened on 27 February 2012. The last participant observation occurred on 10 December 2013.
Pre-assignment Details: Part A: 52 participants were screened; 38 were enrolled and treated, and comprise the Part A Safety Analysis Set (SAS) and Part A Full Analysis Set (FAS).
  Part B: 42 participants were screened; 23 were enrolled and treated (9 from Part A and 14 who joined the study), and comprise the Part B SAS and Part B FAS.
Groups:
- Part A: SOF+EFV/FTC/TDF (Cohort 1): Sofosbuvir (SOF; 1 × 400 mg tablet or 2 × 200 mg tablets) + efavirenz (EFV) 600 mg/emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg tablet coadministered once daily for 7 days followed by EFV/FTC/TDF (600/200/300 mg) tablet once daily for 7 days.
- Part A: SOF+EFV+ZDV/3TC (Cohort 2): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + EFV 600 mg tablet once daily + zidovudine (ZDV) 300 mg/lamivudine (3TC) 150 mg tablet twice daily for 7 days followed by EFV 600 mg tablet once daily + ZDV/3TC (300/150 mg) tablet twice daily for 7 days.
- Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + atazanavir (ATV) 400 mg tablet boosted with ritonavir (RTV) 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days followed by ATV 400 mg tablet + RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days.
- Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + darunavir (DRV; 800 mg; 2 × 400 mg tablets) boosted with RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days followed by DRV (800 mg; 2 x 400 mg tablets) + RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days.
- Part A: SOF+RAL+FTC/TDF (Cohort 5): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + raltegravir (RAL) 400 mg tablet twice daily + FTC/TDF (200/300 mg) tablet once daily for 7 days followed by RAL 400 mg twice daily + FTC/TDF (200/300 mg) tablet once daily for 7 days.
- Part B: SOF+PEG+RBV: SOF 400 mg tablet once daily + pegylated interferon alpha (PEG) 180 μg subcutaneous injection once weekly + weight-based ribavirin (RBV; 1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks.
Period: Part A
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5) | Part B: SOF+PEG+RBV
Started | 12 | 4 | 8 | 7 | 7 | 0
Completed | 11 (3 participants from this group continued in the Part B: SOF+PEG+RBV group.) | 4 (No participants from this group continued in the Part B: SOF+PEG+RBV group.) | 8 (3 participants from this group continued in the Part B: SOF+PEG+RBV group.) | 7 (2 participants from this group continued in the Part B: SOF+PEG+RBV group.) | 7 (1 participant from this group continued in the Part B: SOF+PEG+RBV group.) | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5) | Part B: SOF+PEG+RBV
Started | 0 | 0 | 0 | 0 | 0 | 23 (9 participants in this group transferred from a Part A cohort, and 14 participants joined the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 19
Not Completed | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who enrolled and received at least one dose of study drug(s)
Groups:
- Part A: SOF+EFV/FTC/TDF (Cohort 1): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) + EFV/FTC/TDF (600/200/300 mg) tablet coadministered once daily for 7 days followed by EFV/FTC/TDF (600/200/300 mg) tablet once daily for 7 days.
- Part A: SOF+EFV+ZDV/3TC (Cohort 2): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + EFV 600 mg tablet once daily + ZDV/3TC (300/150 mg) tablet twice daily for 7 days followed by EFV 600 mg tablet once daily + ZDV/3TC (300/150 mg) tablet twice daily for 7 days.
- Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + ATV 400 mg tablet boosted with RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days followed by ATV 400 mg tablet + RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days.
- Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + DRV (800 mg; 2 × 400 mg tablets) boosted with RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days followed by DRV (800 mg; 2 x 400 mg tablets) + RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet coadministered once daily for 7 days.
- Part A: SOF+RAL+FTC/TDF (Cohort 5): SOF (1 × 400 mg tablet or 2 × 200 mg tablets) once daily + RAL 400 mg tablet twice daily + FTC/TDF (200/300 mg) tablet once daily for 7 days followed by RAL 400 mg twice daily + FTC/TDF (200/300 mg) tablet once daily for 7 days.
- Part B: SOF+PEG+RBV: SOF 400 mg tablet once daily + PEG 180 μg subcutaneous injection once weekly + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks.
  This reporting group presents data for those participants who joined the study for Part B only.
- Total: Total of all reporting groups
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5) | Part B: SOF+PEG+RBV | Total
Number analyzed (Participants) | 12 | 4 | 8 | 7 | 7 | 14 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.1) | 58 (5.3) | 47 (6.4) | 47 (3.8) | 46 (10.3) | 46 (8.7) | 47 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 1 | 1 | 3 | 8
  Male | 10 | 4 | 7 | 6 | 6 | 11 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 4 | 7 | 7 | 7 | 14 | 51
  Not Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 8 | 2 | 4 | 3 | 7 | 11 | 35
  Black or African American | 4 | 2 | 4 | 4 | 0 | 3 | 17
HCV Genotype [Number; unit: participants] — There are variations of HCV which are all similar enough to be called HCV, but are distinct enough to be referred to as HCV genotypes.
  participants
    Genotype 1A | 5 | 1 | 5 | 5 | 6 | 9 | 31
    Genotype 1B | 5 | 1 | 1 | 0 | 0 | 2 | 9
    Genotype 2B | 1 | 1 | 2 | 0 | 0 | 0 | 4
    Genotype 3A | 0 | 1 | 0 | 2 | 1 | 2 | 6
    Genotype 4 | 1 | 0 | 0 | 0 | 0 | 0 | 1
    Genotype 4A/4C/4D | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A: Plasma Pharmacokinetics of SOF, EFV, Tenofovir (TFV), and FTC: AUCtau at Day 7
Description: AUCtau: concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval).
  Data for this outcome measure were collected for participants in Part A only.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
Population: Pharmacokinetics (PK) Analysis Set: participants with evaluable PK profiles who enrolled into Part A of the study and received study drug.
  Participants in the PK Analysis Set with available data were included.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5)
Number analyzed (Participants) | 8 | 4 | 8 | 7 | 7
h*ng/mL
  Pharmacokinetics of SOF (AUCtau at Day 7) | 867.5 (460.34) | 627.6 (315.87) | 2269.4 (567.58) | 1421.5 (415.10) | 1687.1 (573.42)
  Pharmacokinetics of EFV (AUCtau at Day 7) | 95094.4 (71267.91) | 53770.7 (39263.90) | NA (NA) — No data: EFV was not administered to this group. | NA (NA) — No data: EFV was not administered to this group. | NA (NA) — No data: EFV was not administered to this group.
  Pharmacokinetics of TFV (AUCtau at Day 7) | 2351.2 (960.74) | NA (NA) — No data: TFV was not administered to this group. | 3793.0 (835.11) | 3996.8 (1665.17) | 2657.1 (751.31)
  Pharmacokinetics of FTC (AUCtau at Day 7) | 10144.8 (2832.23) | NA (NA) — No data: FTC was not administered to this group. | 11564.9 (1739.26) | 13091.2 (4093.09) | 10622.8 (815.24)

2. Primary Outcome: Part A: Plasma Pharmacokinetics of SOF, EFV, TFV, and FTC: Cmax at Day 7
Description: Cmax: maximum observed concentration of drug in plasma.
  Data for this outcome measure were collected for participants in Part A only.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 hours postdose
Population: Participants in the PK Analysis Set with available data were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5)
Number analyzed (Participants) | 8 | 4 | 8 | 7 | 7
ng/mL
  Pharmacokinetics of SOF (Cmax at Day 7) | 635.0 (344.19) | 285.1 (62.28) | 1228.9 (474.93) | 828.2 (351.41) | 1189.2 (483.83)
  Pharmacokinetics of EFV (Cmax at Day 7) | 5423.8 (3283.86) | 3469.5 (1707.54) | NA (NA) — No data: EFV was not administered to this group. | NA (NA) — No data: EFV was not administered to this group. | NA (NA) — No data: EFV was not administered to this group.
  Pharmacokinetics of TFV (Cmax at Day 7) | 372.5 (208.71) | NA (NA) — No data: TFV was not administered to this group. | 519.8 (119.89) | 441.8 (134.13) | 388.1 (118.53)
  Pharmacokinetics of FTC (Cmax at Day 7) | 1533.1 (829.88) | NA (NA) — No data: FTC was not administered to this group. | 1797.9 (232.54) | 1808.2 (530.10) | 2079.5 (434.32)

3. Primary Outcome: Part B: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
  Data for this outcome measure were collected for participants in Part B only.
Time Frame: Posttreatment Week 12
Population: Part B Full Analysis Set: participants enrolled into Part B of the study and dosed with at least 1 dose of study drug(s)
Measure: Number; unit: percentage of participants
Groups:
- Part B: SOF+PEG+RBV: SOF 400 mg tablet once daily + PEG 180 μg subcutaneous injection once weekly + weight-based RBV (1000-1200 mg as 200 mg tablets in a divided daily dose) for 12 weeks.
Arm/Group | Part B: SOF+PEG+RBV
Number analyzed (Participants) | 23
percentage of participants | 91.3

4. Secondary Outcome: Part B: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 was defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
  Data for this outcome measure were collected for participants in Part B only.
Time Frame: Posttreatment Weeks 4 and 24
Population: Part B Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part B: SOF+PEG+RBV
Number analyzed (Participants) | 23
percentage of participants
  SVR4 | 91.3
  SVR24 | 91.3

5. Secondary Outcome: Part B: Percentage of Participants Experiencing Viral Breakthrough or Viral Relapse
Description: Viral breakthrough was defined as having confirmed detectable HCV RNA levels (HCV RNA > LLOQ) on treatment after having previously had undetectable HCV RNA levels (HCV RNA < LLOQ) while on treatment.
  Viral relapse was defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) at end of treatment, but did not achieve an SVR.
  Data for this outcome measure were collected for participants in Part B only.
Time Frame: Posttreatment Weeks 4 and 24
Population: Part B Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Part B: SOF+PEG+RBV
Number analyzed (Participants) | 23
percentage of participants
  Viral breakthrough | 0
  Viral relapse | 8.7

6. Other Pre Specified Outcome: Part B: On-treatment HCV RNA
Description: Data for this outcome measure were collected for participants in Part B only.
Time Frame: Up to 8 weeks
Population: Part B Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Part B: SOF+PEG+RBV
Number analyzed (Participants) | 23
log10 IU/mL
  Baseline (n = 23) | 6.59 (0.872)
  Week 1 (n = 20) | 1.65 (0.425)
  Week 2 (n = 22) | 1.38 (0.000)
  Week 4 (n = 23) | 1.38 (0.000)
  Week 6 (n = 23) | 1.38 (0.000)
  Week 8 (n = 21) | 1.38 (0.000)

7. Other Pre Specified Outcome: Part B: On-treatment HIV RNA
Description: Data for this outcome measure were collected for participants in Part B only.
Time Frame: Up to 8 weeks
Population: Part B Safety Analysis Set: participants enrolled in Part B and received at least one dose of study drug(s).
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Part B: SOF+PEG+RBV
Number analyzed (Participants) | 23
copies/mL
  Baseline (n = 23) | 25 (16.4)
  Week 1 (n = 20) | 20 (4.1)
  Week 2 (n = 22) | 20 (3.0)
  Week 4 (n = 22) | 19 (0.0)
  Week 6 (n = 22) | 19 (0.0)
  Week 8 (n = 21) | 19 (0.0)

8. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who received at least 1 dose of study drug(s)
Measure: Number; unit: percentage of participants
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5) | Part B: SOF+PEG+RBV
Number analyzed (Participants) | 8 | 4 | 8 | 7 | 7 | 23
percentage of participants | 0 | 0 | 0 | 0 | 0 | 8.7

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Nine participants from Part A also enrolled into Part B and are included twice for adverse events.
Arm/Group | Part A: SOF+EFV/FTC/TDF (Cohort 1) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) | Part A: SOF+RAL+FTC/TDF (Cohort 5) | Part B: SOF+PEG+RBV
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/8 | 0/7 | 0/7 | 0/23
Other Adverse Events (participants affected / at risk) | 2/12 | 0/4 | 0/8 | 2/7 | 1/7 | 16/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SOF+EFV/FTC/TDF (Cohort 1) (N=12) | Part A: SOF+EFV+ZDV/3TC (Cohort 2) (N=4) | Part A: SOF+RTV+ATV+FTC/TDF (Cohort 3) (N=8) | Part A: SOF+RTV+DRV+FTC/TDF (Cohort 4) (N=7) | Part A: SOF+RAL+FTC/TDF (Cohort 5) (N=7) | Part B: SOF+PEG+RBV (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 12
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 4
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Body temperature decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years